CLINICAL TRIAL: NCT06411509
Title: An Integration of Tai Chi and rTMS for Physical and Psychological Well-being in Older Adults With Sleep Disturbance
Brief Title: Integration of Tai Chi and Repetitive Transcranial Magnetic Stimulation for Sleep Disturbance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Proferssor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V2024-TMS; 1.51.56.BBCN (Other Grant/Funding Number: PolyU Research Centre for Chinese Medicine Innovation)
Record Dates: First submitted 2024-05-04; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Sleep Disturbance; Interaction
MeSH Terms: conditions — Parasomnias | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TC plus active rTMS (Experimental)
  Interventions: Other: TC plus active rTMS
- TC plus sham rTMS (Sham Comparator)
  Interventions: Other: Tai Chi plus sham rTMS
- TC-alone (Experimental)
  Interventions: Behavioral: TC-alone
- Low-intensity physical exercise (Active Comparator)
  Interventions: Behavioral: Low intensity physical exercise

INTERVENTIONS:
Other: TC plus active rTMS — The rTMS intervention is performed using a MagPro X100 by MagVenture with a water-cooled figure-of-eight coil. Before the treatment session, the resting motor threshold of the left abductor pollicis brevis is determined. The rMT is defined as the minimum intensity which produces five motor evoked potential responses of at least 50 μV in 10 trials at rest. A protocol of 1 Hz rTMS at 80% of RMT is applied over the frontal area of the right DLPFC. The coil position is localized using a frameless stereotactic neuronavigation system (TMS-Navigator, Localite GmbH, Bonn, Germany). Participants receive only three sessions of TC per week without rTMS during in the week 1 and 2, and the TC potocol is same as the TC-alone group. Participants receive daily rTMS (30 minutes) for 5 days a week combined with three sessions of TC in the last 2 weeks. Active rTMS deliveres at 1 Hz for 30 min (1800 pulses per session) with the intensity of 80% rMT.
  Arms: TC plus active rTMS
Other: Tai Chi plus sham rTMS — Sham rTMS is administrated the same procedures as the active rTMS but with low intensity of 20% rMT to elicit similar skin sensations and sounds. The TC protocol in this group is the same as the TC-alone group.
  Arms: TC plus sham rTMS
Behavioral: TC-alone — Participants in the TC-alone group attend a simplified Yang style 8-Form Easy TC training program in a group format. Each session lasts for 60 minutes and are conducted three times per week over a period of four weeks. In the first session, the certified TC instructor explains the exercise theory and procedures. The remaining sessions includes 5 to 10 minutes warm-up and a review of TC principles, 45 minutes meditative movements, and 5 to 10 minutes cool-down
  Arms: TC-alone
Behavioral: Low intensity physical exercise — To achieve the same exercise volume with TC-alone group, participants in the low-intensity physical exercise control group attend a four-week exercise training in group format. Exercise sessions are 60 minutes with three times per week. Each exercise session consists of 5 to 10 minutes warm-up, 45 minutes of aerobic training, and a 5 to 10 minutes cool-down.
  Arms: Low-intensity physical exercise

SUMMARY:
This is a novel and the first study to investigate the impacts of the integrated treatment of Tai Chi (TC) and repetitive transcranial magnetic stimulation (rTMS) on sleep disturbances and the potential mechanisms of arousal system. To validate the combination of TC and rTMS as a promising approach for managing sleep disturbance in older adults, the investigators will conduct a four-arm, parallel-group, randomized controlled trial comprising a 4-week treatment phase and a 3-month follow up period. A total of 152 eligible participants will be recruited and randomly assign to the TC plus active rTMS (38 participants), TC plus sham rTMS (38 participants), TC-alone (38 participants), and low-intensity PE (38 participants) control group within two weeks after the baseline assessment. TC plus active rTMS, TC plus sham rTMS, and TC-alone will be compared with a low-intensity PE control group on insomnia severity, various sleep parameters assessed by self-report sleep diary and ActiGraph, emotional states, and physical and mental health related quality of life. The investigators have formulated two hypotheses in this study. First, the three intervention groups, relative to participants undergoing PE, will confer greater improvement in all measured outcomes at post-intervention (T1) and three-month follow-up (T2); and second, in the double-blinded groups, the TC plus active rTMS will show greater improvement in all measured outcomes than TC plus sham rTMS at T1 and T2.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 60 years
2. Active sleep disturbance as indicated by the Pittsburgh Sleep Quality Index (PSQI) score exceeding 5 and the Insomnia Severity Index (ISI) score greater than 7 at screening
3. No prior experience of mind-body exercises (i.e., TC, Qigong, or yoga, etc.) and regular moderate-intensity exercise (i.e., above three times per week and 30 minutes per session) in the past 6 months
4. Provide written informed consent

Exclusion Criteria:

1. Cognitive impairment as determined by the Montreal Cognitive Assessment scored less than 22
2. Major confounding conditions known to induce sleep perturbations, such as psychiatric disorders or chronic pain disorder
3. History of head injury or epilepsy, intracranial implant, cardiac pacemaker, or any other contraindication to rTMS
4. Obvious physical disability that precluded participant in the interventions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Measured by Insomnia Severity Index, it's a 7-item questionnaire assessing insomnia severity over the past two weeks. Items scored 0 to 4 and total score range is from 0 to 28. Total score of 7 or less indicate no clinically significant insomnia, 8 to 14 indicate subthreshold insomnia, and 15 or greater indicate moderate to severe insomnia.

SECONDARY OUTCOMES:
Actigraphy-assessed sleep parameters | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Collected from a wrist ActiGraph wGT3X-BT on the nondominant hand for 7 consecutive days.
Self-reported sleep parameters | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Derived from a consensus sleep diary for 7 days
Daytime sleepiness | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Evaluated by the Epworth sleepiness scale (ESS). The ESS is used to rate the possibility to doze off or fall asleep. Items scored 0 to 3 and the sum ranges from 0 to 24. The total score exceeds 10 suggests signifies pathological sleepiness, and higher values reflects greater severity.
Emotional states | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Measured by Depression, Anxiety, and Stress Scale-21 Items. Each subscale has seven items that are scored on a 4-point Likert scale (0=not at all to 3=most of the time). More severe symptoms are indicated by higher scores.
Mental function and physical function | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  The self-reported quality of life is measured by the Short Form 36-item Health Survey (SF-36) (Brazier et al. 1992). In the SF-36, the data are presented as physical component score (PCS) and mental component score (MCS). Each domain is valued from 0 to 100, with higher score denoting better health status.
Somatic arousal and cognitive arousal | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  Somatic arousal and cognitive arousal are assessed by the the Pre-Sleep Arousal Scale (PSAS). The PSAS is a 16-item self-reported questionnaire that assesses the state of arousal when falling asleep and is composed of somatic and cognitive arousal subscales with eight items in each. The somatic subscale (PSAS somatic) contains items addressing physical arousal such as racing heart, muscle tension, and rapid breathing. The cognitive subscale (PSAS cognitive) contains items on the worry about falling asleep, being mentally alert at bedtime, and the inability to shut off one's thoughts. Each subscale item is scored on a scale from 1 (not at all) to 5 (extremely). Total scores for each of the subscales can range from 8 to 40, with higher scores associated with greater arousal.
Cortical arousal | at Week 0 (baseline), Week 4 (posttreatment), and Week 16 (follow-up)
  EEG data are collected using the DSI-24 wearable EEG device for 5 minutes in the resting state with eyes closed. Spectral power analysis and functional connectivity analysis will be conducted. Participants with lower cortical arousal shows a decrease in beta- and gamma-band power during the wakefulness eye-closed resting state. In addition, decreased connectivity in the default mode network and increased connectivity in fronto-parietal network is also suggested the improvements of cortical arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Tsang, Professor, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Department of Rehabilitation Sciences, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR